CLINICAL TRIAL: NCT01700504
Title: Effect of Gentamicin Lavage of the Axillary Surgical Bed After Lymph Node Dissection on Drainage Discharge Volume
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Associate Professor Universidad Miguel Hernandez, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012/0009
Record Dates: First submitted 2012-09-24; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Axillary Drainage Volume After Lymph Node Dissection.
Keywords: Axillary drainage volume; Lavage with gentamicin solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Gentamicin lavage (Experimental): Patients undergoing an axillary lavage with 500ml of normal saline followed by 500ml gentamicin solution
  Interventions: Drug: Axillary lavage with gentamicin solution
- Normal saline lavage (Active Comparator): Patients undergoing 2 axillary lavages with 500ml of normal saline
  Interventions: Drug: Axillary lavage with gentamicin solution

INTERVENTIONS:
Drug: Axillary lavage with gentamicin solution — Patients undergoing an axillary lavage with 500ml of normal saline followed by 500ml gentamicin solution

SUMMARY:
The effect of axillary lavage with a gentamicin solution before wound closure will reduce the drainage volume and subsequently day of drainage removal.

DETAILED DESCRIPTION:
Inclusion criteria will be a diagnosis of mammary neoplasms and plans to undergo an elective ALND of Berg´s levels I and II due to axillary metastasis determined preoperatively by core biopsy or evidence of metastasis in the SLNB in the intraoperative or in the differed analysis. Exclusion criteria will be chronic renal failure due to possible toxicity of gentamicin and patients undergoing a modified radical mastectomy.

The patients will be randomized by means of an Internet randomization module into 2 groups: those patients undergoing 2 lavages of the axillary surgical bed with normal saline (Group 1) and those ones first undergoing lavage with normal saline followed by a second lavage with a gentamicin solution (Group 2).

Surgical dissection will be performed using harmonic scalpel (Ultracision, Ethicon Endosurgery, Johnson and Johnson, Cincinnati, OH, USA). Once finished the ALND, a Jackson-Pratt drain will be left in place and connected to a low pressure vacuum device.

Methodology: Irrigation technique and extraction of microbiological samples:

The lavage will be performed immediately prior to closure of the wound, once placed the drainage into the cavity. In both groups, prior to the lavage, a microbiological sample from the surgical bed will be obtained with a swab (sample 1), followed by a lavage with 500 ml normal saline. After aspiration of the saline, a new microbiological sample will be obtained (sample 2). In Group 1 a second lavage with 500 ml normal saline will be performed, while in Group 2 the second lavage will be performed with an antibiotic solution, including gentamicin (240 mg) dissolved in 500 ml normal saline. After aspirating this second lavage, a third microbiological sample will be obtained in the same way as the two previous ones, in both groups (sample 3).

Indication of drain removal and obtention of sample 4:

After discharge, the patient will be asked to quantify the drainage volume daily. Drain will be removed when drainage volume was <30 ml/day. The drainage volume of the last day was collected in a syringe for microbiological study (sample 4).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mammary neoplasms and plans to undergo an elective ALND of Berg´s levels I and II due to axillary metastasis determined preoperatively by core biopsy or evidence of metastasis in the SLNB in the intraoperative or in the differed analysis.

Exclusion Criteria:

* chronic renal failure due to possible toxicity of gentamicin
* patients undergoing a modified radical mastectomy.

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Drainage volume | 7 days
  The drainage volumen between groups (interventional and control)will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Elche, Elche, Alicante, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Cansado P, Perez-Soler M, Gomez MA, Llavero C, Calero P, Zubiaga L, Diez M, Arroyo A, Calpena R. Effect of gentamicin lavage of the axillary surgical bed after lymph node dissection on drainage discharge volume. Breast. 2013 Oct;22(5):874-8. doi: 10.1016/j.breast.2013.03.008. Epub 2013 Apr 18. PMID 23602424